CLINICAL TRIAL: NCT02008526
Title: Theory-based Text Messaging to Reduce Methamphetamine Use and HIV Risks Among MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA035092 (NIH)
Record Dates: First submitted 2013-12-03; First posted 2013-12-11 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-06

CONDITIONS: Methamphetamine Abuse; HIV
Keywords: Text Messaging; mHealth; Methamphetamine; HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TXT-PHE (Experimental): Gay-specific, Theory-based Text Messages Transmitted by Peer Health Educators (TXT-PHE)
  This condition is interactive and tailored to the needs of the individual participant. PHEs initiate (i.e., "push") text messages to participants and also respond to participant-initiated queries and participant responses to the PHE messages (i.e., "pull").
  Participants receive five pre-written messages per day sent on a predetermined schedule. Participants who respond to the pre-written text messages or initiate queries or requests for support ("pull") are sent additional real-time messages back from the PHE.
  During the 8-week intervention, participants receive a brief weekly text-based assessment on their methamphetamine use and HIV sexual behaviors in the previous seven days.
  Interventions: Behavioral: Text Messages Transmitted by Peer Health Educators (TXT-PHE)
- TXT-Auto (Experimental): Group 2: Gay-specific, Theory-based Text Messages Transmitted by Automation (TXT-Auto)
  Participants assigned to this group receive automatic text-messages.
  Following the initial welcome message, participants receive five pre-written messages per day sent on a predetermined schedule.
  During the 8-week intervention, participants receive a brief weekly text-based assessment on their methamphetamine use and HIV sexual behaviors in the previous seven days.
  Interventions: Behavioral: Text Messages Transmitted by Automation (TXT-Auto)
- Assessment Only (AO) (No Intervention): During the 8-week intervention, participants receive a brief weekly text-based assessment on their methamphetamine use and HIV sexual behaviors in the previous seven days.

INTERVENTIONS:
Behavioral: Text Messages Transmitted by Peer Health Educators (TXT-PHE) — Participants receive five gay-specific, theory-based pre-written messages per day sent on a predetermined schedule. Participants who respond to the pre-written text messages or initiate queries or requests for support ("pull") are sent additional real-time messages back from the PHE. Text messages are transmitted and responded to in real time, at the peak hours of high-risk activities. During the 8-week intervention, participants receive a brief weekly text-based assessment on their methamphetamine use and HIV sexual behaviors in the previous seven days.
  Arms: TXT-PHE
Behavioral: Text Messages Transmitted by Automation (TXT-Auto) — Participants receive five gay-specific, theory-based pre-written messages per day sent on a predetermined schedule. During the 8-week intervention, participants receive a brief weekly text-based assessment on their methamphetamine use and HIV sexual behaviors in the previous seven days.
  Arms: TXT-Auto

SUMMARY:
Participants receive culturally relevant and specifically tailored text messages based on the behavioral change theoretical constructs of Social Support Theory, Health Belief Model, and Social Cognitive Theory. Participants are randomized into one of three conditions for an 8-week intervention period: Group 1: culturally relevant theory-based text messages interactively transmitted by peer health educators (TXT-PHE); or, Group 2: the same culturally relevant theory-based text messages transmitted by automation (TXT-Auto); or, Group 3: assessment-only (AO) control with no theoretically based text messages.

DETAILED DESCRIPTION:
The randomized three-group design uses repeated assessments at baseline, at the end of the 8-week intervention period, and at 3-, 6-, and 9-month post randomization follow-up. Participants in all three conditions receive brief weekly text-message assessments on their methamphetamine use and HIV sexual behaviors in the previous seven days. This study will determine the differential immediate and sustained effects of transmitting theory-based text messages by PHE (TXT-PHE) versus by automation (TXT-Auto), compared to an assessment-only (AO) control condition among out-of-treatment, methamphetamine-using MSM for reductions of methamphetamine use and HIV sexual risk behaviors. It is hypothesized that there will be significantly greater reductions in methamphetamine use and HIV sexual risk behaviors from text messages transmitted by PHE than by text messages transmitted by automation, which in turn will produce significantly greater reductions than the AO condition (PHE > TXT > AO). In addition, this study will determine the cost-effectiveness of TXT-PHE vs. TXT-Auto compared to AO for reducing methamphetamine use and HIV sexual risk behaviors. The investigators hypothesize that the TXT-PHE intervention will prove more cost-effective than TXT-Auto in reducing methamphetamine use and HIV sexual risk behaviors, while the TXT-Auto condition will prove more cost effective than the AO condition in reducing these same outcomes (PHE > TXT > AO).

ELIGIBILITY:
Inclusion Criteria:

* Self-identified MSM
* Between the ages of 18 and 65 years
* Methamphetamine use within the previous 3 months
* Unprotected anal intercourse (insertive or receptive) with a non-primary male partner in the previous 6 months
* Not currently in treatment or seeking methamphetamine abuse treatment
* Able and willing to fully charge a cellular phone daily
* Able and willing to provide informed consent
* Able and willing to comply with study requirements

Exclusion Criteria:

* Does not identify as a MSM
* Not between the ages of 18 and 65 years
* Has not used methamphetamine in the previous 3 months
* Has not had unprotected anal intercourse (insertive or receptive) with a non-primary male partner in the previous 6 months
* Currently in treatment or seeking methamphetamine abuse treatment
* Unable or unwilling to fully charge a cellular phone daily
* Unable or unwilling to provide informed consent
* Unable or unwilling to comply with study requirements
* Unable to understand the Informed Consent Form
* Determined to have a more serious psychiatric condition (SCID verified) that is beyond the safe enrollment of study procedures

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy J Reback, Ph.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Community Center, a division of Friends Research Institute, Inc., Los Angeles, CA 90028, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reback CJ, Ling D, Shoptaw S, Rohde J. Developing a Text Messaging Risk Reduction Intervention for Methamphetamine-Using MSM: Research Note. Open AIDS J. 2010 May 14;4:116-22. doi: 10.2174/1874613601004030116. PMID 20657827
- [Background] Reback CJ, Grant DL, Fletcher JB, Branson CM, Shoptaw S, Bowers JR, Charania M, Mansergh G. Text messaging reduces HIV risk behaviors among methamphetamine-using men who have sex with men. AIDS Behav. 2012 Oct;16(7):1993-2002. doi: 10.1007/s10461-012-0200-7. PMID 22610370

RESULTS

PARTICIPANT FLOW:
Groups:
- TXT-PHE: Gay-specific, Theory-based Text Messages Transmitted by Peer Health Educators (TXT-PHE)
  Interactive and tailored to the needs of the individual participant. PHEs initiate text messages to participants and also respond to participant-initiated queries and participant responses to the PHE messages.
  Participants receive five pre-written messages per day. Participants who respond to the pre-written text messages or initiate queries or requests for support are sent additional messages back.
  During the 8-week intervention, participants receive a brief weekly text-based assessment on their methamphetamine use and HIV sexual behaviors in the previous seven days.
  Text Messages Transmitted by Peer Health Educators (TXT-PHE): Text messages are transmitted and responded to in real time, at the peak hours of high-risk activities. Participants receive a brief weekly text-based assessment on their methamphetamine use and HIV sexual behaviors in the previous seven days.
- TXT-Auto: Group 2: Gay-specific, Theory-based Text Messages Transmitted by Automation (TXT-Auto)
  Participants assigned to this group receive automatic text-messages.
  Following the initial welcome message, participants receive five pre-written messages per day sent on a predetermined schedule.
  During the 8-week intervention, participants receive a brief weekly text-based assessment on their methamphetamine use and HIV sexual behaviors in the previous seven days.
  Text Messages Transmitted by Automation (TXT-Auto): Participants receive five gay-specific, theory-based pre-written messages per day sent on a predetermined schedule. During the 8-week intervention, participants receive a brief weekly text-based assessment on their methamphetamine use and HIV sexual behaviors in the previous seven days.
Period: Overall Study
Arm/Group | TXT-PHE | TXT-Auto | Assessment Only (AO)
Started | 94 | 99 | 93
Completed | 86 | 85 | 84
Not Completed | 8 | 14 | 9
Not completed — Death | 0 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 2
Not completed — Lost to Follow-up | 5 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TXT-PHE | TXT-Auto | Assessment Only (AO) | Total
Number analyzed (Participants) | 94 | 99 | 93 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.04 (11.31) | 41.00 (11.12) | 41.43 (10.15) | 41.48 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 94 | 99 | 93 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 29 | 23 | 72
  Not Hispanic or Latino | 74 | 70 | 70 | 214
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 40 | 45 | 40 | 125
  White | 20 | 16 | 20 | 56
  More than one race | 10 | 6 | 6 | 22
  Unknown or Not Reported | 21 | 29 | 25 | 75
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 94 | 99 | 93 | 286
HIV Status [Count of Participants; unit: Participants]
  HIV Negative | 57 | 57 | 54 | 168
  HIV Positive | 37 | 42 | 39 | 118

OUTCOME MEASURES:

1. Primary Outcome: Methamphetamine Use
Description: Self-reported and/or biomarker-confirmed methamphetamine use assessed at baseline and 9-month follow-up assessment.
Time Frame: 9-months post randomization
Population: Number of participants retained through 9-month follow-up.
Measure: Mean (Standard Deviation); unit: Days Used in the Past 30 Days
Arm/Group | TXT-PHE | TXT-Auto | Assessment Only (AO)
Number analyzed (Participants) | 94 | 99 | 93
Days Used in the Past 30 Days
  Baseline Meth Use | 11.13 (9.53) | 10.75 (9.48) | 10.34 (9.00)
  9-Month Follow-up Meth Use: number analyzed (Participants) | 86 | 85 | 84
  9-Month Follow-up Meth Use | 7.79 (9.83) | 7.05 (9.87) | 5.66 (7.89)
Statistical Analysis 1: Comparison: TXT-PHE vs TXT-Auto vs Assessment Only (AO); Test type: Superiority; p = 0.3137, ANOVA; 2 Degrees of Freedom; F = 1.16

2. Primary Outcome: HIV Sexual Risk Behavior
Description: Engagement in condomless anal intercourse was assessed at baseline and 9-month post-randomization follow-up.
Time Frame: 9-months post randomization
Population: Participants retained through nine months post randomization.
Measure: Mean (Standard Deviation); unit: # Episodes (Past 30 Days)
Arm/Group | TXT-PHE | TXT-Auto | Assessment Only (AO)
Number analyzed (Participants) | 94 | 99 | 93
# Episodes (Past 30 Days)
  Baseline Condomless Anal Intercourse | 11.44 (15.58) | 14.05 (19.49) | 7.39 (12.91)
  9-Month Follow-up Condomless Anal Intercourse: number analyzed (Participants) | 86 | 85 | 84
  9-Month Follow-up Condomless Anal Intercourse | 5.19 (12.84) | 4.34 (11.56) | 4.31 (9.41)
Statistical Analysis 1: Comparison: TXT-PHE vs TXT-Auto vs Assessment Only (AO); Test type: Superiority; p = 0.8494, ANOVA; 2 Degrees of Freedom; F = 0.16

3. Primary Outcome: Cost Effectiveness
Description: Cost-effectiveness data is collected quarterly throughout the course of the study using the UNAIDS template.
Time Frame: up to 36 months
Reporting Status: Not Posted

4. Secondary Outcome: HIV Primary Care
Description: HIV-positive participants will be assessed according to their linkage/retention in HIV primary care and adherence to ART medication at 8-weeks, 3-, 6-, and 9-months post-randomization.
Time Frame: 8-weeks post randomization, 3-/6-/9-months post randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For up to 9-months post randomization
Arm/Group | TXT-PHE | TXT-Auto | Assessment Only (AO)
All-Cause Mortality (participants affected / at risk) | 0/94 | 2/99 | 1/93
Serious Adverse Events (participants affected / at risk) | 0/94 | 2/99 | 1/93
Other Adverse Events (participants affected / at risk) | 0/94 | 0/99 | 0/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TXT-PHE (N=94) | TXT-Auto (N=99) | Assessment Only (AO) (N=93)
Death (General disorders) | 0 (0) | 2 (2) | 1 (1) — Participant death.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes